CLINICAL TRIAL: NCT01854788
Title: A Comparative Study of Three Airway Clearance Techniques With Different Autonomy Degrees in Non Cystic Fibrosis Bronchiectasis: Randomized Cross-over Trial.
Brief Title: 3 Airway Clearance Techniques in Non Cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Beatriz Herrero, Physiotherapist, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Uniko2010.01
Record Dates: First submitted 2012-08-08; First posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Bronchiectasis
Keywords: Airway clearance techniques; Mucus clearance; Chest physiotherapy; Autogenic drainage; Slow expiration with glottis opened in lateral posture(ELTGOL); Temporary-positive expiratory pressure (T-PEP); Non cystic fibrosis bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Autogenic drainage (Active Comparator): All patients performed all interventions in a randomized order. Each technique was applied in 3 non consecutively sessions during one week. The time spent during the session was 40 minutes
  Interventions: Other: Autogenic drainage
- Slow expiration with glottis opened in lateral posture (Active Comparator): All patients performed all interventions in a randomized order.Each technique was applied in 3 non consecutively sessions during one week. The time spent during the session was 40 minutes
  Interventions: Other: Slow expiration with glottis opened in lateral posture
- Temporary-Positive Expiratory Pressure (Active Comparator): All patients performed all interventions in a randomized order. Each technique was applied in 3 non consecutively sessions during one week. The time spent during the session was 40 minutes
  Interventions: Other: Temporary-positive expiratory pressure

INTERVENTIONS:
Other: Autogenic drainage — It was performed following J. Chevallier recommendations.In this trial it was considered a self-administrated technique because physiotherapist only gave oral advice in order to ensure a correct performance of the technique.
  Arms: Autogenic drainage
Other: Slow expiration with glottis opened in lateral posture — It was performed following Postiaux´s recommendations. In this trial the technique was considered active-assisted because the physiotherapy played a role important in their execution.
  Other Names: Slow expiratory with glotis opened in lateral position
  Arms: Slow expiration with glottis opened in lateral posture
Other: Temporary-positive expiratory pressure — The diaphragmatic breathing was required for this technique whereas patients remain seated in front of the device with a nose clip. The inspiratory /expiratory ratio was 1:2.It was taken into account as a device-administrated technique for this trial.
  Arms: Temporary-Positive Expiratory Pressure

SUMMARY:
Study design: a randomized, crossover trial. Each patient performed three different airway clearance techniques (Autogenic drainage, slow expiratory with glottis opened in lateral posture [ELTGOL], temporary- positive expiratory pressure [T-PEP] with not similar autonomy degree in a randomized order. Each technique were applied in 3 sessions during one week at alternate days (Monday /Wednesday/Friday or Tuesday/Thursday/Saturday). The time spent in each bronchial session was 40 minutes. Seven days were the wash-out time period between the different techniques.

ELIGIBILITY:
Inclusion Criteria:

1. - Non Cystic Fibrosis bronchiectasis diagnosed by High Resolution Computed Tomographic
2. - Mean sputum production ≥ 15 ml /24h
3. - Clinical stability in the last 6 weeks
4. - Not carrying out regular chest physiotherapy
5. - Forced expiratory volume in 1 second ≥ 30% pred. ; Forced Vital Capacity ≥ 45% pred. and peak expiratory flow >270 L/s

Exclusion Criteria:

1. - Smoker or non-smoker form less than 2 years
2. - Cystic fibrosis
3. - Active tuberculosis or sarcoidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Weight of sputum expectorated during each airway clearance therapy session | 40 minutes
  Wet weight sputum production were recollected in one pre-weighted containers. It was measured in grams.
Weight of sputum expectorated 24 hours post each bronchial session | 24 hours
  Wet weight sputum production were recollected in one pre-weighted containers. It was measured in grams.

SECONDARY OUTCOMES:
Saint George Respiratory Questionnaire (SGRQ) | Change from baseline at 5 weeks
  Saint George Respiratory Questionnaire (SGRQ) is a self-completed health-related quality of life questionnaire.It was validated in bronchiectasis. It was administrated at the start and at the end of trial.
Leicester Cough Questionnaire (LCQ) | Changes from baseline arm to 1 week
  Leicester Cough Questionnaire is a self-completed quality of life measure of the impact of cough severity. It was validated in bronchiectasis. It was administrated at the start and at the end of each technique.

OTHER OUTCOMES:
Lung function measured by simple spirometry: forced expiratory volume in 1 second, Forced vital capacity, Forced expiratory flow 25-75 | Change from baseline arm to 1 week
Likert test | Change from baseline arm to 1 week
  It is a patient´s preferences measure. The questionnaire consists of a package of simple questions about the airway clearance techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Herrero, Phy, Principal Investigator — Hospital Clinic of Barcelona; Eva Polverino, Doctor, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital CLinic, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Herrero-Cortina B, Alcaraz-Serrano V, Torres A, Polverino E. Reliability and Minimum Important Difference of Sputum Weight in Bronchiectasis. Respir Care. 2020 Oct;65(10):1478-1487. doi: 10.4187/respcare.07175. Epub 2020 Feb 18. PMID 32071136
- [Derived] Herrero-Cortina B, Vilaro J, Marti D, Torres A, San Miguel-Pagola M, Alcaraz V, Polverino E. Short-term effects of three slow expiratory airway clearance techniques in patients with bronchiectasis: a randomised crossover trial. Physiotherapy. 2016 Dec;102(4):357-364. doi: 10.1016/j.physio.2015.07.005. Epub 2015 Dec 1. PMID 26712530